CLINICAL TRIAL: NCT06370754
Title: A Phase Ib/II Platform Trial of Newly Emerging Immunotherapy for Pancreatic Cancer Treatment
Brief Title: Newly Emerging Immunotherapy for Pancreatic Cancer Treatment
Acronym: FD-IMPACT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, M.D.,Ph.D., Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2401289-19-2403
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — toripalimab; irinotecan sucrosofate; Fluorouracil; Leucovorin; Taxes; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort1: JS004+JS001+Irinotecan Liposome Injection+5-fluorouracil (5-FU)/leucovorin (LV) (Experimental): Participants with unresectable locally advanced or metastatic pancreatic cancer who had previously failed at least first line gemcitabine-based system therapy will receive JS004 and JS001 combined with chemotherapy (irinotecan liposome injection+5-FU/LV) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS004; Drug: Irinotecan Liposome Injection; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)
- Cohort2: JS007+JS001+Irinotecan Liposome Injection+5-FU/LV (Experimental): Participants with unresectable locally advanced or metastatic pancreatic cancer who had previously failed at least first line gemcitabine-based system therapy will receive JS007 and JS001 combined with chemotherapy (irinotecan liposome injection+5-FU/LV) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS007; Drug: Irinotecan Liposome Injection; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)
- Cohort3: JS015+JS001+Irinotecan Liposome Injection+5-FU/LV (Experimental): Participants with unresectable locally advanced or metastatic pancreatic cancer who had previously failed at least first line gemcitabine-based system therapy will receive JS015 and JS001 combined with chemotherapy (irinotecan liposome injection+5-FU/LV) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS015; Drug: Irinotecan Liposome Injection; Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin (LV)
- Cohort4: JS004+JS001+Nab-Paclitaxel+Gemcitabine (Experimental): Participants with previously untreated systemic pancreatic cancer with unresectable locally advanced or metastatic pancreatic cancer will receive JS004 and JS001 combined with chemotherapy (nab-paclitaxel+gemcitabine) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS004; Drug: Nab paclitaxel; Drug: Gemcitabine
- Cohort5: JS007+JS001+Nab-Paclitaxel+Gemcitabine (Experimental): Participants with previously untreated systemic pancreatic cancer with unresectable locally advanced or metastatic pancreatic cancer will receive JS007 and JS001 combined with chemotherapy (nab-paclitaxel+gemcitabine) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS007; Drug: Nab paclitaxel; Drug: Gemcitabine
- Cohort6: JS015+JS001+ Nab-Paclitaxel+Gemcitabine (Experimental): Participants with previously untreated systemic pancreatic cancer with unresectable locally advanced or metastatic pancreatic cancer will receive JS015 and JS001 combined with chemotherapy (nab-paclitaxel+gemcitabine) until the treatment termination event specified in the protocol occurs.
  Interventions: Drug: JS001; Drug: JS015; Drug: Nab paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: JS001 — 240 mg by IV infusionevery 3 weeks (Q3W), given on cycle day 1.
  Other Names: Toripalimab
Drug: JS004 — 200 mg by IV infusion Q3W, given on cycle day 1.
  Arms: Cohort1: JS004+JS001+Irinotecan Liposome Injection+5-fluorouracil (5-FU)/leucovorin (LV); Cohort4: JS004+JS001+Nab-Paclitaxel+Gemcitabine
Drug: JS007 — 3mg/kg by IV infusion Q3W, given on cycle day 1.
  Arms: Cohort2: JS007+JS001+Irinotecan Liposome Injection+5-FU/LV; Cohort5: JS007+JS001+Nab-Paclitaxel+Gemcitabine
Drug: JS015 — 600mg by IV infusion Q3W, given on cycle day 1.
  Arms: Cohort3: JS015+JS001+Irinotecan Liposome Injection+5-FU/LV; Cohort6: JS015+JS001+ Nab-Paclitaxel+Gemcitabine
Drug: Irinotecan Liposome Injection — 60 or 70 mg/m^2 by IV infusion every 2 weeks (Q2W), given on cycle day 1.
  Arms: Cohort1: JS004+JS001+Irinotecan Liposome Injection+5-fluorouracil (5-FU)/leucovorin (LV); Cohort2: JS007+JS001+Irinotecan Liposome Injection+5-FU/LV; Cohort3: JS015+JS001+Irinotecan Liposome Injection+5-FU/LV
Drug: 5-Fluorouracil (5-FU) — 2400mg/m^2, intravenously, over 46 h on day 1, Q2W.
  Arms: Cohort1: JS004+JS001+Irinotecan Liposome Injection+5-fluorouracil (5-FU)/leucovorin (LV); Cohort2: JS007+JS001+Irinotecan Liposome Injection+5-FU/LV; Cohort3: JS015+JS001+Irinotecan Liposome Injection+5-FU/LV
Drug: Leucovorin (LV) — 400mg/m^2, intravenously, over 30 min on day 1, Q2W.
  Arms: Cohort1: JS004+JS001+Irinotecan Liposome Injection+5-fluorouracil (5-FU)/leucovorin (LV); Cohort2: JS007+JS001+Irinotecan Liposome Injection+5-FU/LV; Cohort3: JS015+JS001+Irinotecan Liposome Injection+5-FU/LV
Drug: Nab paclitaxel — 125 mg/m^2 by IV infusion Q3W, given on cycle day 1 and 8.
  Arms: Cohort4: JS004+JS001+Nab-Paclitaxel+Gemcitabine; Cohort5: JS007+JS001+Nab-Paclitaxel+Gemcitabine; Cohort6: JS015+JS001+ Nab-Paclitaxel+Gemcitabine
Drug: Gemcitabine — 1000 mg/m^2 by IV infusion Q3W, given on cycle day 1 and 8.
  Arms: Cohort4: JS004+JS001+Nab-Paclitaxel+Gemcitabine; Cohort5: JS007+JS001+Nab-Paclitaxel+Gemcitabine; Cohort6: JS015+JS001+ Nab-Paclitaxel+Gemcitabine

SUMMARY:
This is a Phase Ib/II platform clinical study to evaluate the initial efficacy and safety of different novel immunotherapies in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
The cohort A/B/C included patients with unresectable locally advanced or metastatic pancreatic cancer who had previously failed at least first line gemcitabine-based system therapy.The cohort D/E/F included patients with previously untreated systemic pancreatic cancer with unresectable locally advanced or metastatic pancreatic cancer.This study plans to first explore A/B/C cohort, and then start the D/E/F cohort after determining the safety.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation, written informed consent, complied well and cooperated with the follow-up visits;
* Age ≥ 18 years old, female or male individuals;
* Eastern Cooperative Oncology Group (ECOG) Performance status score of 0 or 1, the expected survival is more than 3 months;
* Patients with locally advanced unresectable or metastatic pancreatic cancer confirmed by histopathology or cytopathology (islet cell tumor is not eligible for inclusion) who meet the following requirements:

  * For the A/B/C/ cohort: Had failed of at least first-line systemic therapy; disease recurrence or progression within 6 months of the last treatment of neoadjuvant or adjuvant chemotherapy was also allowed to be enrolled;
  * For the D/E/F cohort: No prior systemic treatment; patients with recurrence or progression of disease more than 6 months after the last treatment of neoadjuvant or adjuvant chemotherapy were also allowed to be enrolled;
* Had at least one measurable lesion according to RECIST v1.1.
* Patients had adequate major organs function;
* Women of childbearing potential must undergo serum pregnancy test within 7 days prior to the first dose and the result must be negative. Female subjects of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 180 days after the last dose of study drug.

Exclusion Criteria:

* Previously received drugs with the same target as the planned investigational therapy;
* radiotherapy (except for palliative reasons), endocrine therapy, chemotherapy, immunotherapy, or molecular targeted therapy within 4 weeks prior to initial administration, except for bisphosphonates (which can be used for bone metastasis);
* Uncontrolled central nervous system metastases (meaning symptoms or the use of glucocorticoids or mannitol to control symptoms);
* A history of clinically significant or uncontrolled heart disease, including congestive heart failure, angina pectoris, myocardial infarction, or ventricular arrhythmia, in the 6 months prior to initial dosing;
* Patients with Grade 1 and above adverse reactions caused by previous treatment, including Grade 1 peripheral neurotoxicity; hair loss is not included and the investigator should clearly record the reasons;
* Malignant tumors within 5 years prior to the first dose (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
* Active autoimmune disease requiring systemic treatment within 2 years prior to first administration, except for vitiligo, type I diabetes, residual hypothyroidism due to autoimmune thyroiditis requiring hormone replacement therapy only;
* History of rapid allergic reaction, eczema or asthma that cannot be controlled by topical corticosteroids;
* Patients who have lung disease, such as drug-induced interstitial lung disease or pneumonia, obstructive pulmonary disease that severely affects lung function, and symptomatic bronchospasm;
* Serious infections requiring antibiotic treatment within 14 days prior to initial administration (>CTCAE grade 2), such as severe pneumonia, bacteremia, comorbidifications, etc., resulting in the need for hospitalization;
* Vaccination of live vaccine within 4 weeks before the first dose or during the study period;
* Known human immunodeficiency virus (HIV) infection, allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* History of prior allergy to any component or excipient of the investigational drug to be received;
* Other conditions assessed by the investigator as unsuitable for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) (phase IB) | 21 days after the first dose was administered to each subject
  If less than 2 participants developed DLT during the safety observation period (one cycle after the first dose), follow-up first-line D/E/F cohort exploration should be considered. Otherwise, it is up to the investigator to decide the next research plan.
Objective Response Rate (ORR) (phase II) | Up to 1 year
  ORR was defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR) based on RECIST 1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (phase IB) | Up to 1 year
  ORR was defined as the percentage of participants with a best overall response of CR or PR based on RECIST 1.1.
Disease control rate (DCR) | Up to 1 year
  DCR was defined as the percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable based on RECIST 1.1.
Duration of Response (DOR) | Up to 1 year
  DOR will be calculated from the date of the first evaluation showing PR, or CR, to the date of the first disease progression or death, whichever comes first and based on RECIST 1.1.
Progression free survival (PFS) | Up to 2 years
  PFS is defined as the time from the first dose until objective tumor progression(PD), or death, whichever comes first and based on RECIST 1.1. At the end of the study, the time of last acquisition of living patients without PD was taken as the deleted data.
Overall Survival (OS) | Up to 2 years
  OS will be measured from the date of first dose to death from any cause.
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 90 days after the last administration
  Adverse event (AE), abnormal laboratory examination, serious adverse event (SAE) related with the study drug judged using NCI-CTCAE V5.0 by investigator.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China